CLINICAL TRIAL: NCT00709956
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Crossover Study to Assess the Effects of a Single Dose of Iloprost Power 15 on Exercise Capacity in Patients With Symptomatic Pulmonary Arterial Hypertension
Brief Title: Iloprost Power 15 in Pulmonary Arterial Hypertension
Acronym: PROWESS 15
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-063A301
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Ventavis; iloprost; inhaled treatment; pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active / placebo (Experimental): Single dose of iloprost (5 µg) on study day 2 followed by single dose of placebo on study day 3
  Interventions: Drug: iloprost (5 µg); Drug: placebo
- Placebo / active (Placebo Comparator): Single dose of placebo on study day 2 followed by single dose of iloprost (5 µg) on study day 3
  Interventions: Drug: iloprost (5 µg); Drug: placebo

INTERVENTIONS:
Drug: iloprost (5 µg) — Single dose of iloprost 5 µg using I-neb(R) Adaptive Aerosol Delivery (AAD(R)) System power setting 15 disc
  Other Names: Ventavis(R)
Drug: placebo — Single dose of matching placebo using I-neb(R) Adaptive Aerosol Delivery (AAD(R)) System power setting 15 disc

SUMMARY:
Patients with symptomatic idiopathic pulmonary arterial hypertension (IPAH), or familial pulmonary arterial hypertension (FPAH) or pulmonary hypertension associated with Human immunodeficiency virus (HIV) or drugs/toxins in New York Heart Association (NYHA) functional class II to IV at baseline, naive to PAH treatment or currently being treated with a stable dose of either bosentan, ambrisentan or sildenafil will be enrolled in the PROWESS 15 study. This randomized, double blind, placebo-controlled, crossover, and single-dose study will determine whether a single inhaled dose of iloprost using the power 15 disc improves exercise capacity compared to placebo in patients with pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study mandated procedure,
* Patients with symptomatic idiopathic, or familial pulmonary arterial hypertension or pulmonary hypertension associated with human immunodeficiency virus (HIV) or drugs/toxins in NYHA functional class II to IV.
* Women of childbearing potential must have a negative urine pregnancy test and must use an adequate method of contraception during the study and for 28 days after discontinuation of the study drug.

Exclusion Criteria:

* Pulmonary arterial hypertension related to any condition other than those specified in the inclusion criteria,
* Pulmonary arterial hypertension associated with significant venous or capillary involvement (Pulmonary capillary wedge pressure (PCWP) > 15 mmHg),
* Known pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis,
* Moderate to severe obstructive lung disease: forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 65% of predicted value after bronchodilator administration,
* Moderate to severe restrictive lung disease: total lung capacity (TLC) < 60% of predicted value,
* Pregnant or breast-feeding women,
* Systemic hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg on repeated measurement),
* Systolic blood pressure < 95 mmHg,
* Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C,
* Chronic renal insufficiency defined by serum creatinine > 2.5 mg/dL (221 μmol/L) or ongoing dialysis,
* Clinically relevant bleeding disorder or active bleeding,
* For those patients on monotherapy, any contraindication to bosentan, ambrisentan, or sildenafil, according to product label,
* Known hypersensitivity to iloprost or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laila Rouault, MD, Study Director — Actelion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: On Day 1 all patients received a single inhalation dose of placebo. Patients who satisfied the selection criteria in the single-blind period of the study were entered into the double-blind period to receive iloprost 5 μg and matching placebo (Days 2 and 3) in a single dose, two-period crossover design.
Pre-assignment Details: Of the 70 randomized patients, 64 patients entered the double-blind period, (placebo/iloprost P15, 33 patients and iloprost P15/placebo, 31 patients). 1 patient in the iloprost P15/placebo treatment sequence was excluded from the per-protocol analysis which was defined as the primary analysis.
Groups:
- Iloprost (5µg) / Placebo: Single dose double-blind active iloprost (5µg) on study day 2 followed by single dose double-blind placebo on study day 3
- Placebo / Iloprost (5 µg): Single dose double-blind placebo on study day 2 followed by single dose double-blind active iloprost (5µg) on study day 3
Period: Overall Study
Arm/Group | Iloprost (5µg) / Placebo | Placebo / Iloprost (5 µg)
Started | 33 (Day 1 Single-blind placebo run-in) | 37 (Day 1 Single-blind placebo run-in)
Double-blind Crossover-period | 31 (Days 2 and 3) | 33 (Days 2 and 3)
Completed | 30 | 33
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Inclusion/exclusion criteria violation | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloprost (5µg) / Placebo | Placebo / Iloprost (5 µg) | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 46
  >=65 years | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (13.57) | 55.8 (16.40) | 55.7 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 28 | 30 | 58
  Austria | 2 | 2 | 4
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: 6-minute-walk Distance (6MWD)
Description: The 6-minute walk test was performed 20-40 minutes after treatment. This was a non-encouraged test (the person conducting the test did not encourage the patient to walk farther or faster) that measured the distance covered over a 6-minute walk.
  It was conducted by a trained member of the site staff who was listed on the site's delegation of authority sheet. For patients who had never performed a 6-minute walk test previously, a training test was requested before the qualifying tests for randomization.
Time Frame: Study day 2 or study day 3
Population: The analysis was per protocol, 64 patients started double blind phase of study, 63 completed.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | 6MWD After Placebo Treatment | 6MWD After Iloprost (5 µg) Treatment
Number analyzed (Participants) | 63 | 63
meters | 330.0 (22.84) [322.3 to 337.7] | 328.6 (55.28) [320.9 to 336.2]
Statistical Analysis 1: Comparison: 6MWD After Placebo Treatment vs 6MWD After Iloprost (5 µg) Treatment; With a sample size of at least 63 patients and based on the assumptions on the primary endpoint (normal distribution, SD of the difference of 30 m) the study was designed to detect a significant treatment effect with 90% power, assuming a difference exceeding 12.5 m between the mean values of the 6MWD following the iloprost power 15 treatment and the one following the placebo treatment; Test type: Superiority or Other; p = 0.7883, Generalized linear model — If the primary endpoint reaches significance, treatment effect of the secondary endpoint is determined at a 2-sided nominal of 0.05. Since hierarchy of the endpoints to be tested has been predefined, no correction for multiple testing will be applied; Subject (sequence), treatment, and period as fixed effect; Difference in least squares mean = -1.5, 95% CI 2-sided [-12.3 to 9.4]

2. Secondary Outcome: Borg Dyspnea Score
Description: The Borg scale is a category-ratio scale, commonly used to evaluate the effects of exercise on dyspnea. The original and modified scales have ratio properties ranging from 0 = nothing at all to 10 = very, very severe, with descriptors from 0 to 10. Descriptors have been modified by others so that 10 has been labeled "extremely severe," or "the worst possible dyspnea imaginable." Reliability and validity have been reported in a general population and in patients with PAH as well as other respiratory conditions.
Time Frame: Study day 2 or study day 3
Population: The analysis was per protocol, 64 patients started double blind phase of study, 63 completed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Borg Dyspnea Score After Placebo Treatment | Borg Dyspnea Score After Iloprost (5 µg) Treatment
Number analyzed (Participants) | 63 | 63
scores on a scale | 3.5 (2.23) | 3.4 (2.25)

ADVERSE EVENTS:
Description: Due to data capture design constraints the time of adverse event (AE) onset was not collected, therefore the potential to assign potential causality to active treatment or placebo was not assessed. AE's can only be reported as shown, as prospectively planned in the protocol submitted to FDA. Includes all patients entered in the double-blind phase.
Arm/Group | Iloprost (5µg) / Placebo | Placebo / Iloprost (5 µg)
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/33
Other Adverse Events (participants affected / at risk) | 16/31 | 20/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iloprost (5µg) / Placebo (N=31) | Placebo / Iloprost (5 µg) (N=33)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost (5µg) / Placebo (N=31) | Placebo / Iloprost (5 µg) (N=33)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Flushing (Vascular disorders) | 4 | 5
Headache (Nervous system disorders) | 3 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No